CLINICAL TRIAL: NCT03769883
Title: The Effects of Different Doses of Exercise on Pancreatic ß-cell Function in Patients With Newly Diagnosed Type 2 Diabetes (DOSE-EX): A Randomized Clinical Trial
Brief Title: Exercise Volume and Beta-cell Function in T2D The DOSE-EX Randomized Trial
Acronym: DOSE-EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathias Ried-Larsen (Other)
Responsible Party: Sponsor-Investigator, Mathias Ried-Larsen, Principal investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-18038298
Record Dates: First submitted 2018-11-22; First posted 2018-12-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus; Type2 Diabetes; Diabetes Mellitus, Type 2; Type2 Diabetes Mellitus
Keywords: Exercise; Physical Activity; Type 2 diabetes; Pancreatic beta-cell function; Insulin sensitivity; Dose finding; lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Insulin Resistance | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Upon completion of the study and prior to breaking the allocation code, a data-collection form is generated by a statistician and the principal investigator. The data-analyst breaks the allocation code and labels the participants according to the assigned treatment and analyzes the outcomes. Following the analyses, group allocation will be concealed in all data outputs and the N per group and present the data to the writing committee in a blinded fashion. Then the writing committee will provide their blinded interpretations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary control (DCON) (Experimental): The macro-nutrient distributions are in line with the current guidelines from the national Diabetes Association and Canadian guidelines, where individualization in macronutrient distribution should lie within the range of 45-60E% carbohydrate, 15-20E% protein and 20-35E% fat. The dietary plan will aim at reducing saturated fat intake <7E% aiming at a caloric deficit of 500 kilo calories/day
  Interventions: Behavioral: Diet
- Moderate Exercise Dose (MED) (Experimental): Two aerobic training sessions per week of 45-60 min duration and one session per week with combined aerobic (30-35 min) and resistance (30 min) training and a dietary intervention (as above)
  Interventions: Behavioral: Exercise and diet
- High Exercise Dose (HED) (Experimental): Four aerobic training sessions per week of 45-60 min duration and two sessions per week with combined aerobic (30-35 min) and resistance (30 min) training and a dietary intervention (as above)
  Interventions: Behavioral: Exercise and diet
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Exercise and diet — The participants will undergo diet or combined diet and exercise. The exercise will be provided at different volumes
  Arms: High Exercise Dose (HED); Moderate Exercise Dose (MED)
Behavioral: Diet — Dietary intervention
  Arms: Dietary control (DCON)

SUMMARY:
This project will provide an exercise-based lifestyle intervention with the potential to reduce complications for patients with short standing type 2 diabetes (T2D). While exercise is widely accepted as a component of T2D management, little is known about the additive effect of exercise when combined with a diet on T2D pathophysiology and mechanisms believed to lead to micro- and macrovascular complications. Moreover, the necessary dose of exercise to revert the progression of T2D and the related complications has not been investigated. A large-scale randomized controlled trial (RCT) will be essential to document the effectiveness on reducing the risk of T2D complications. However, prior to conducting a large-scale RCT, we need to specify the exercise dose that efficiently compliments the diet.

In a 4-armed randomized, clinical trial (N=80 T2D patients, T2D duration < than 7 years) we aim to investigate 1) the potential additive role of exercise on pancreatic β-cell function in patients with T2D when combined with a diet, 2) the causal relationship between lifestyle-induced reductions in glycaemic variability, oxidative stress and low-grade inflammation and, 3) the role of exercise in rescuing dysregulated muscle progenitor cells. The participants will be randomly allocated to either a) control, b) diet, c) diet and exercise 3 times/week or d) diet and exercise 6 times/week for 16 weeks. Prior to, during and following the interventions, all participants will undergo extensive testing.

DETAILED DESCRIPTION:
A 4-armed, 16-week, parallel-group, assessor-blinded, randomized, clinical trial. Participants will be randomly allocated (1:1:1:1), stratified by sex

Interventions:

The lifestyle interventions will consist of two main components; 1) increased physical activity and structured exercise and/or 2) a dietary intervention aiming at a weight loss. Whereas there will be no differences in the dietary intervention between the lifestyle groups, the volume of physical activity and structured exercise will vary according to the frequencies of the structured exercise sessions.

The study groups are prescribed:

1. Control group (CON): No intervention
2. Dietary control (DCON): Dietary intervention (see below)
3. Moderate Exercise Dose (MED): Two aerobic training sessions per week of 45-60 min duration and one session per week with combined aerobic (30-35 min) and resistance (30 min) training and a dietary intervention (described below)
4. High Exercise Dose (HED): Four aerobic training sessions per week of 45-60 min duration and two sessions per week with combined aerobic (30-35 min) and resistance (30 min) training and a dietary intervention (described below)

Detailed description of the intervention components. Exercise: The training protocol will be adapted based on a previous study where the T2D participants were prescribed 6 weekly sessions of aerobic training alone or combined aerobic and resistance training (averaging 360-420 min of exercise per week). As previous analyses suggest that there may be an inverse dose-response relationship between reductions in HbA1c and aerobic exercise volume, this parameter will be used to adapt the training protocol. As the effect of exercise on HbA1c is closer related to the number of training sessions rather than intensity15, we will reduce the number of sessions by 50%, to three sessions/week in the moderate exercise dose group and maintain the original session frequency in the high dose exercise group (six sessions/week).Training will be supervised and monitored to ensure intensity and compliance.

Dietary intervention and intended weight loss (DCON, MED and HED: The dietary intervention will be based on the recommendations from the American Diabetes Association (ADA) with increased focus on macronutrient quality. The macronutrient distributions are in line with the current guidelines from the national Diabetes Association and Canadian guidelines, where individualization in macronutrient distribution should lie within the range of 45-60 energy% carbohydrate, 15-20 energy% protein and 20-35 energy% fat. Thus, the dietary intervention emphasis will be on low glycemic index and low glycemic load in shape of non-processed foods and will aim at reducing saturated fat intake <7 energy%.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with diabetes type 2 and/or HbA1c ≥ 48 mmol/mol if no treatment with anti-diabetic medication and/or use of antidiabetic medication

Caucasian

No diagnose of Type 1 diabetes, mature onset diabetes of the young, Latent autoimmune diabetes of adults

T2D 0-6 years of duration

No treatment with insulin

Body Mass Index (BMI) >27 kg/m2 and <40 kg/m2

No known or signs of intermediate or severe microvascular complications to diabetes (retino-, neuro- or nephropathy)

No known cancer

No Known lung disease

No known cardiovascular disease

No known thyroid disease

No known liver disease

No known autoimmune disease

No other endocrine disorder causing obesity

No current treatment with anti-obesity medication

No current treatment with anti-inflammatory medication

No weight loss of > 5kg within the last 6 months

No diagnose of depression or treatment with anti-depressive medication, ongoing or within the last three months before enrolment

No diagnose of psychiatric disorder or treatment with anti-psychotic medication

No history of suicidal behavior or ideations within the last three months before enrolment

No previous surgical treatment for obesity (excluding liposuction > 1 year prior to enrolment)

Not pregnant/considering pregnancy

No functional impairments that prevents the performance of intensive exercise

Accept of medical regulation by the U-TURN endocrinologist

Inactivity, defined as < 1,5 hours of structured physical activity pr. week at moderate intensity and cycling < 30 minutes/5 km pr. day at moderate intensity (moderate intensity = out of breath but able to speak)

No participation in other research intervention studies

Exclusion Criteria:

HbA1c: >=75 mmol/mol with no glucose lowering medications

HbA1c: >=64 mmol/mol with mono glucose lowering therapy (if compliant with the prescription)

HbA1c: >=57 mmol/mol with >=dual glucose lowering therapy (if compliant with the prescription)

estimated glomerular filtration rate<60 mL/min

Protein or glucose in the urine at pre-screening

No biochemical sign of other major diseases

Presence of circulating glutamate-decarboxylase anti body (GAD) 65

Objective findings that contraindicates participation in intensive exercise

Anamnestic findings that contraindicates participation in the study

Unable to allocate the needed time to fulfill the intervention

Language barrier, mental incapacity, unwillingness or inability to understand and be able to complete the interventions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Pancreatic beta-cell function (Per protocol) | From baseline (0 weeks) to follow-up (16 weeks)
  The change in the late-phase disposition index (DI) during the final 30 minutes of hyperglycemic phase of the hyperglycemic clamp.

SECONDARY OUTCOMES:
Pancreatic beta-cell function (Intention to treat) | From baseline (0 weeks) to follow-up (16 weeks)
  As for per protocol
Glucagon like peptide 1 sensitivity (c-peptide) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Glucagon like peptide 1 stimulated C-peptide secretion
Glucagon like peptide 1 sensitivity (glucagon) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Glucagon like peptide 1 stimulated glucagon secretion
Glucagon like peptide 1 sensitivity (insulin) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Glucagon like peptide 1 stimulated insulin secretion
Arginine sensitivity (insulin) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Arginine stimulated insulin secretion
Arginine sensitivity (c-peptide) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Arginine stimulated C-peptide secretion
Arginine sensitivity (glucagon) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Arginine stimulated glucagon secretion
Early phase disposition index (c-peptide) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in 1st phase C-peptide secretion defined as the peak concentration during the initial 10 minutes of the hyperglycaemic clamp
Early phase disposition index (insulin) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in 1st phase insulin secretion defined as the peak concentration during the initial 10 minutes of the hyperglycaemic clamp
Glucose clearance | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Rate of glucose clearance (stable isotope infusion) during steady state hyperglycemia
Glucose appearance | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Rate of glucose appearance (stable isotope infusion) during steady state hyperglycemia
Insulin sensitivity | From baseline (0 weeks) to follow-up (16 weeks)
  Change in mean Glucose infusion rate over last 30 min of clamp phase/(mean insulin×glucose
Mean amplitude of glycemic excursions | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Mean amplitude of glycemic excursions (MAGE - calculated based on min 3 days sensor glucose profiles)
Coefficient of glucose variation | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Coefficient of variation defined as (mean glucose/the standard deviation (SD)) of min 3 days sensor glucose profiles
Mean glucose levels | From baseline (0 weeks) to follow-up (16 weeks)
  Change in the mean glucose levels (calculated based on min 3 days sensor glucose profiles)
Time in hyperglycemia | From baseline (0 weeks) to follow-up (16 weeks)
  Change in time in hyperglycaemia (calculated based on min 3 days sensor glucose profiles)
Time in hypoglycemia | From baseline (0 weeks) to follow-up (16 weeks)
  Change in time in hypoglycaemia from min 3 days sensor glucose profiles
Pancreatic fat | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Pancreatic fat
Hepatic fat | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Hepatic fat
Visceral fat | From baseline (0 weeks) to follow-up (16 weeks)
  Change in visceral fat
Total fat mass | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Total fat mass
Total fat free mass | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Total fat free mass
Total lean body mass | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Total lean body mass
Android fat mass | From baseline (0 weeks) to follow-up (16 weeks)
  Change in Android fat mass
Gynoid fat mass | From baseline (0 weeks) to follow-up (16 weeks)
  Change in gynoid fat mass
Body weight | From baseline (0 weeks) to follow-up (16 weeks)
  Change in body weight
Body mass index | From baseline (0 weeks) to follow-up (16 weeks)
  Change in body mass index
Systemic oxidative stress (RNA) | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in 8-oxo-guanosine
Systemic oxidative stress (DNA) | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in 8-oxo-deoxoguonase
Advanced glycation end-products (AGE) | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in AGE
The circulating receptor for advanced glycation end-products (sRAGE) | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in sRAGE
Markers of low-grade inflammation | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in inflammatory markers (e.g. high sensitive C-reactive protein, interferon-ϒ, interleukin-10, interleukin-8, interleukin-6, interleukin-1, TNFα)
Glycated haemoglobin type 1AC (HbA1c) | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in HbA1c
Total cholesterol | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in total cholesterol
Total triglyceride | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in total triglyceride
Low density lipoprotein (LDL) | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in LDL
High density lipoprotein (HDL) | From baseline (0 weeks) to follow-up (4, 12 and 16 weeks)
  Change in HDL
Systolic blood pressure | From baseline (0 weeks) to follow-up (16 weeks)
  Change systolic blood pressures
Diastolic blood pressure | From baseline (0 weeks) to follow-up (16 weeks)
  Change diastolic blood pressure
Glucose tolerance | From baseline (0 weeks) to follow-up (16 weeks)
  Change incremental and total area under the curve (glucose, c-peptide, insulin) during a mixed meal tolerance test
Gastric emptying (AUC) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in the AUC (paracetamol) during a mixed meal tolerance test
Gastric emptying (Rate of appearance) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in rate of appearance of paracetamol during a mixed meal tolerance test
Physical fitness (VO2max) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in physical fitness (VO2) during a progressive maximal bicycle ergometer test
Muscular 1 repetition max (strength) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in 1 repetition max
Total physical activity | From baseline (0 weeks) to follow-up (16 weeks)
  Change in objectively measured physical activity (counts per minute)
Moderate and vigorous physical activity (MVPA) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in time spend on MVPA
Sedentary time (SED) | From baseline (0 weeks) to follow-up (16 weeks)
  Change in time spend on SED
Physical well being | From baseline (0 weeks) to follow-up (16 weeks)
  Change in physical well being (Based on the physical dimension score from short-form 36, range 0-100)
Mental well being | From baseline (0 weeks) to follow-up (16 weeks)
  Change in mental well being (Based on the mental dimension score from Short-form 36) (range 0-100)
Satiety | From baseline (0 weeks) to follow-up (16 weeks)
  Change in self-reported satiety (VAS) during a mixed meal tolerance test (range 0-10)

OTHER OUTCOMES:
Muscular metabolic function | From baseline (0 weeks) to follow-up (16 weeks)
  Change in metabolic function (Based on muscle biopsies in a subset of participants, N=16-32))
Fat tissue metabolic function | From baseline (0 weeks) to follow-up (16 weeks)
  Change in metabolic function (Based on muscle biopsies in a subset of participants, N=16-32)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ried-Larsen, PhD, Principal Investigator — Centre for Physical Activity Research, Righospitalet
Locations (1):
- Center for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
If the data can be fully anonymized the data can be shared.

REFERENCES:
- [Background] Lyngbaek MPP, Legaard GE, Bennetsen SL, Feineis CS, Rasmussen V, Moegelberg N, Brinklov CF, Nielsen AB, Kofoed KS, Lauridsen CA, Ewertsen C, Poulsen HE, Christensen R, Van Hall G, Karstoft K, Solomon TPJ, Ellingsgaard H, Almdal TP, Pedersen BK, Ried-Larsen M. The effects of different doses of exercise on pancreatic beta-cell function in patients with newly diagnosed type 2 diabetes: study protocol for and rationale behind the "DOSE-EX" multi-arm parallel-group randomised clinical trial. Trials. 2021 Apr 1;22(1):244. doi: 10.1186/s13063-021-05207-7. PMID 33794975
- [Result] Legaard GE, Lyngbaek MPP, Almdal TP, Karstoft K, Bennetsen SL, Feineis CS, Nielsen NS, Durrer CG, Liebetrau B, Nystrup U, Ostergaard M, Thomsen K, Trinh B, Solomon TPJ, Van Hall G, Brond JC, Holst JJ, Hartmann B, Christensen R, Pedersen BK, Ried-Larsen M. Effects of different doses of exercise and diet-induced weight loss on beta-cell function in type 2 diabetes (DOSE-EX): a randomized clinical trial. Nat Metab. 2023 May;5(5):880-895. doi: 10.1038/s42255-023-00799-7. Epub 2023 May 1. PMID 37127822
- [Result] Legaard GE, Lyngbaek MPP, Almdal TP, Durrer CG, Nystrup U, Larsen EL, Poulsen HE, Karstoft K, Pedersen BK, Ried-Larsen M. Effects of different doses of exercise in adjunct to diet-induced weight loss on the AGE-RAGE axis in patients with short standing type 2 diabetes: Secondary analysis of the DOSE-EX multi-arm, parallel-group, randomised trial. Free Radic Biol Med. 2023 Nov 1;208:52-61. doi: 10.1016/j.freeradbiomed.2023.07.031. Epub 2023 Jul 31. PMID 37532066